CLINICAL TRIAL: NCT06992232
Title: Radiotherapy or Radical Prostatectomy Combined With Intense Androgen Deprivation Therapy for Newly Diagnosed Metastatic Prostate Cancer: A Multi-center Randomized Controlled Phase II Trial
Brief Title: Radiotherapy or Surgery Combined With Intense Androgen Deprivation Therapy for mCRPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); Peking University First Hospital, Beijing, CHINA (Unknown)
Responsible Party: Principal Investigator, Hongqian Guo, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-122
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer Metastatic Disease
Keywords: metastatic prostate cancer; radiotherapy; prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intense androgen deprivation therapy (IADT) (Active Comparator): Patients received ADT plus ARi (enzalutamide, apalutamide, darolutamide or rezvilutamide) for 2 years in the Intense androgen deprivation therapy (IADT) group.
  Interventions: Drug: Intense androgen deprivation therapy
- Radiotherapy or Surgery plus IADT (Experimental): For patients in the experimental group, local treatment either radiotherapy or surgery was arranged in addition to systemic ADT plus ARi. Those allocated radiotherapy received 70Gy/2.8Gy/25f schedule for primary tumor and 70Gy/2.6-2.8Gy/25f or 37.5Gy/7.5Gy/5f for metastatic lymph nodes and bone lesions based on the size and location. While those allocated surgery received robot-assisted laparoscopic radical prostaectomy plus extended pelvic lymph node dissection for local treatment.
  Interventions: Drug: Intense androgen deprivation therapy; Radiation: Radiation Therapy; Procedure: radical prostatectomy

INTERVENTIONS:
Drug: Intense androgen deprivation therapy — Patients received ADT plus second-generation ARi (enzalutamide, apalutamide, darolutamide or rezvilutamide) for 2 years.
  Other Names: ADT plus second-generation ARi
Radiation: Radiation Therapy — Those allocated radiotherapy received 70Gy/2.8Gy/25f schedule for primary tumor and 70Gy/2.6-2.8Gy/25f or 37.5Gy/7.5Gy/5f for metastatic lymph nodes and bone lesions based on the size and location. Radiation should be finished within 2 years' systemic therapy.
  Arms: Radiotherapy or Surgery plus IADT
Procedure: radical prostatectomy — Those allocated surgery received robot-assisted laparoscopic radical prostaectomy plus extended pelvic lymph node dissection for local treatment. Surgery should be finished within 2 years' systemic therapy.
  Arms: Radiotherapy or Surgery plus IADT

SUMMARY:
This multi-center randomized controlled phase II trial was carried out in several hospitals in China to evaluate the efficacy and safety of radiotherapy or radical prostatectomy combined with intense androgen deprivation therapy for newly diagnosed metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate adenocarcinoma, with distant metastasis diagnosed by novel imaging modalities (PSMA PET/CT or PSMA PET/MR), involving ≤10 metastatic sites (amenable to local therapy) and without visceral metastasis.
2. The primary lesion is deemed resectable, or can achieve a resectable state following IADT.
3. Non-castration range (≥50 ng/dl), or the duration of testosterone levels in the castration range is no more than 3 months.
4. Eastern Cooperative Oncology Group (ECOG) physical condition score ≤ 1.
5. Patients must have adequate hematologic function, hepatic function and renal function.
6. Patients must participate voluntarily and sign an informed consent form(ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must be willing to obey the prohibitions and restrictions specified in the research protocol.
7. Fertile patients must be willing to use highly effective contraception during the study period.

Exclusion Criteria:

1. Patients with prostatic histopathology exhibiting neuroendocrine, small cell, or sarcomatoid features.
2. The researchers assessed the primary lesion as unresectable.
3. Patients who had previously received androgen deprivation therapy (including medical or surgical castration) for more than 3 months, or had undergone focal therapy for prostate cancer, or had received radiotherapy or chemotherapy for prostate cancer.
4. Patients with severe or uncontrolled underlying diseases who could not tolerate surgery or radiotherapy.
5. Patients with New York Heart Association (NYHA) Class III/IV congestive heart failure, unstable angina, or a history of myocardial infarction within the past 6 months.
6. Uncontrolled severe hypertension, persistently uncontrolled diabetes, oxygen-dependent pulmonary disease, chronic liver disease, or HIV infection.
7. Within the past 5 years, having had other malignant tumors except for prostate cancer, with the exception of cured basal or squamous cell skin cancer.
8. Suffering from mental illness, mental disability, or being incapable of providing informed consent.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival | 2 years
  Following 2 years of treatment, any anti-tumor treatment was terminated for those who met complete remission until two consecutively rised PSA>0.2ng/ml. Complete remission is interpreted as PSA level<0.1ng/ml and absence of radiographic as well as clinical progression following the 2-year treatment, both are indispensable. The primary outcome was event-free survival (EFS), defined as the time from disease complete remission to any required anti-tumor treatment.

SECONDARY OUTCOMES:
progression-free survival | 4 years
  Defined as from treatment initiation to PSA progression or radiographic/clinical progression. PSA progression is defined as PSA >1 ng/ml, with two consecutive PSA measurements at least one week apart showing a 50% or greater increase from baseline). Radiographic progression is defined as development of two or more new bone metastases or progression of soft tissue lesions according to RECIST 1.1 criteria. Clinical progression is defined as worsening clinical symptoms and signs as determined by the physician.
Time to CRPC | 4 years
  Time to CRPC (castration-resistant prostate cancer (CRPC) is calculated from treatment initiation to the development of CRPC. CRPC is defined as serum testosterone at castration level (<50 ng/dl or 1.7 nmol/l), while meeting one of the following criteria: a. Biochemical progression: Three consecutive PSA rises, each measured at least one week apart, with at least two increases exceeding 50% above baseline, and at least one PSA value >2 ng/ml. b. Radiographic progression: Development of two or more new bone metastases, or progression of soft tissue lesions according to RECIST criteria.
Adverse events | 4 years
  valuate all adverse events (AEs) and grade them according to NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR